CLINICAL TRIAL: NCT02645864
Title: Apatinib and Irinotecan Combination as Second-line Treatment in Esophageal Squamous Cell Carcinoma: a Phase I Dose Escalation Study
Brief Title: Apatinib and Irinotecan Combination Treatment in Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaodong Zhang, Doctor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBE001
Record Dates: First submitted 2015-12-23; First posted 2016-01-05 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2017-04

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; Apatinib; Irinotecan
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — apatinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib and Irinotecan (Experimental): This study will include a sequential evaluation of 3 subjects per cohort. Cohort 1: apatinib 250 mg per day and irinotecan 150mg q2w. Cohort 2: apatinib 500 mg per day and irinotecan 150mg q2w. Cohort 3: apatinib 750 mg per day and irinotecan 150mg q2w.
  A dose limiting toxicity (DLT) event is defined as any of the following events:
  * CTCAE Grade 4 event
  * Grade 3 non-hematologic toxicity including fever, nausea, vomiting, and diarrhea that continues despite optimal medical management) If a DLT is experienced in any cohort, the cohort will be expanded to 6 subjects. If two (2) DLTs are experienced in any cohort, the study will stop and the dose of combination treatment in this cohort will be documented.
  Interventions: Drug: Apatinib; Drug: Irinotecan

INTERVENTIONS:
Drug: Apatinib — 250mg p.o. qd in first cohort (3 subjects). 250mg p.o. bid in second cohort (3 subjects) 250mg p.o. tid in third cohort (3 subjects)
  Other Names: YN968D1
Drug: Irinotecan — 150mg/m^2 i.v. q2w
  Other Names: Camptosar, Campto

SUMMARY:
Esophageal cancer is one of the common malignant tumors. The annual incidence of esophageal squamous cell carcinoma is 260,000 with the mortality of 210,000 in China. Different from that in western countries, esophageal squamous cell carcinoma (ESCC) is still the dominant pathological type in China and account for more than 95% cases in clinic. The prognosis of ESCC is very poor. About 50% of patients have advanced disease at diagnosis with a 5-year survival rate of only 5-7%. Though esophagectomy is standard treatment, disease will relapse in many patients.

For patients with unresectable or recurrent disease, chemotherapy is an important treatment alone or with radiotherapy. Taxane, platinum, and fluoropyrimidine have been reported effective in ESCC and is popularly used in first-line treatment of ESCC. However, there is still no standard 2nd-line treatment for patients who fail in first-line treatment. Both irinotecan and taxane had been studied as 2nd-line treatment for esophageal cancer patients. But there are only a few of ESCC patients involved in those studies.

Except for chemotherapy, targeting treatment is another promising treatment for esophageal cancer. In recent years, antiangiogenic treatment has been proved to be effective and tolerable in many cancers such lung, colorectal, and gastric cancer. Apatinib is an also known as YN968D1, is an orally antiangiogenic agents. Preclinical and clinical data has shown that it is effective in the treatment of a variety of solid tumors including esophageal cancer. And it was approved and launched in China in 2014 as a 3rd-line treatment for patients with advanced gastric cancer.

Therefore, investigators initialize this dose escalation phase I study to explore the safety of irinotecan and apatinib combination treatment in ESCC patients with relapse disease after esophagectomy and failure in 1st-line chemotherapy. Investigators will analyze the maximum tolerated dose (MDT) and dose-limiting toxicity (DLT) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed esophageal squamous cell carcinoma with relapse disease and the primary tumor have been surgically removed.

  * With measurable or evaluable disease defined by RECIST 1.1 criteria by multi-slice spiral CT or MRI scan.
  * - Failed in or disease progressed after fist-line chemotherapy (If failed in perioperative chemotherapy or disease progressed in 24 weeks after perioperative chemotherapy, the perioperative chemotherapy is regard as first-line chemotherapy )
  * - Patients must have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale
  * - Without serious system dysfunction and could tolerate chemotherapy.
  * - With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥100g/L (without blood transfusion during 14 days); a neutrophil count of ≥2.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.
  * - Life expectancy ≥3 months
  * - With normal electrocardiogram results and no history of congestive heart failure.
  * - Without bleeding and thrombosis disease
  * - With normal coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT) and INR, each ≤ 1.5 x ULN
  * - Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug
  * - With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
  * - With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

* Patients who have received irinotecan or apatinib in previous treatment.
* Primary tumor is not resected.
* Uncontrolled hypertension (after treatment with antihypertensive drugs cannot reduced to the normal range: systolic pressure <140 mmHg and diastolic pressure <90 mmHg)
* With ≥ grade 2 coronary heart disease, arrhythmia (including corrected QT interval prolongation male >450 ms, women >470 ms)
* Cannot take oral tables including uncontrolled vomiting, chronic diarrhea and intestinal obstruction.
* With potential bleeding risk including (1) peptic ulcer and fecal occult blood (++); (2) melena or hematemesis history in last 3 months; (3) fecal occult blood (+) or (+/-) and endoscopy showed ulcer or other diseases with bleeding risk.
* With abnormal coagulation function (INR>1.5 ULN, APTT>1.5 ULN),
* With thrombosis or receiving anticoagulant treatment.
* With serious diseases such as congestive heart failure, uncontrolled myocardial infarction and arrhythmia, liver failure and renal failure.
* With brain metastasis of tumor
* Pregnant or lactated women (premenopausal women must give urine pregnancy test before enrollment).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | From enrollment to 1 months after completion of treatment. Estimated about 3 months.
  Dose limiting toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 4.0 criteria.
Maximum tolerance dose | From enrollment to 1 months after completion of treatment. Estimated about 3 months.
  Maximum tolerance dose (MTD) is the dose of treatment in the cohort where there are 2 cases of DTL reported.

SECONDARY OUTCOMES:
Objective response rate | From enrollment to 3 months after treatment
  Definition of ORR: clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate).
Progression-free survival | From enrollment to progression of disease. Estimated about 6 months.
  Definition of PFS: The length of time from enrollment until the time of progression of disease (PFS, progression-free survival).
Overall survival | From enrollment to death of patients. Estimated about 1 year.
  Definition of OS: The length of time from enrollment until the time of death (OS, overall survival).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No